CLINICAL TRIAL: NCT02457468
Title: The Coflex®COMMUNITY Study: An Observational Study of Coflex® Interlaminar Technology
Status: Completed | Type: Observational
Sponsor: Predicted, Reported and Observed Outcomes Foundation (Other)
Collaborators: SPIRITT Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: SR-2015-01
Record Dates: First submitted 2015-05-10; First posted 2015-05-29 (Estimated); Last update posted 2019-12-24 (Actual); Status verified 2019-02

CONDITIONS: Spinal Stenosis
Keywords: coflex; interlaminar stabilization; lumbar spinal stenosis; neurogenic claudication; decompression
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stenosis patients treated with coflex: Patients with a primary diagnosis of lumbar spinal stenosis treated with coflex after decompression
  Interventions: Device: coflex

INTERVENTIONS:
Device: coflex

SUMMARY:
The purpose of the coflexCOMMUNITY observational study is to collect information on patients with spinal stenosis undergoing back surgery with the coflex® implant, and to look at their outcomes and the cost-effectiveness of this procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is skeletally mature and has at least moderate impairment in function, experiences relief in flexion from his/her symptoms of leg/buttocks/groin pain, with or without back pain, and has undergone at least 6 months of non-operative treatment;
2. Patient is treated surgically at 1 or 2 contiguous lumbar motion segments with the coflex Interlaminar Device from L1-L5 after decompression of stenosis at the affected level(s), where such use is not contraindicated as noted below.

Exclusion Criteria:

1. Prior fusion or decompressive laminectomy at any index lumbar level;
2. Radiographically compromised vertebral bodies at any lumbar level(s) caused by current or past trauma or tumor (e.g., compression fracture);
3. Severe facet hypertrophy that requires extensive bone removal which would cause instability;
4. Grade II or greater spondylolisthesis;
5. Isthmic spondylolisthesis or spondylolysis (pars fracture);
6. Degenerative lumbar scoliosis (Cobb angle of greater than 25°);
7. Osteoporosis;
8. Back or leg pain of unknown etiology;
9. Axial back pain only, with no leg, buttock, or groin pain;
10. Morbid obesity defined as a body mass index > 40;
11. Active or chronic infection - systemic or local;
12. Known allergy to titanium alloys or magnetic resonance imaging (MRI) contrast agents;
13. Cauda equina syndrome defined as neural compression causing neurogenic bowel or bladder dysfunction;
14. Vulnerable population including pregnant women, prisoners, students and employees of treating physicians, and others who can be subject to coercion;
15. Patient is unwilling to complete his/her surveys.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cohort will be selected from clinic patients scheduled for surgery with coflex device after decompression
Sampling Method: Non-Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2015-06; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Improvement in the Oswestry Disability Index (ODI), compared to pre-surgery | 5 years
  The primary variable of performance is the assessment of Oswestry Low Back Pain Disability Index (ODI). It will be assessed if the improvement in ODI since the pre-surgery status is at least 15 points
Patient has not undergone any reoperations, removals, revisions, or supplemental fixations; | 5 years
  Assessment of reoperations, revisions, removals, or supplemental fixation associated with the coflex device.
Patient has not had any major device related complications | 5 years
  Assessment of major device-related complications, including but not limited to permanent new or increasing sensory or motor deficit at 2 years and 5 years.
Patient has not undergone any Epidural injections | 5 years
  Assessment of lumbar epidural injections

SECONDARY OUTCOMES:
Zurich Claudication Questionnaire (ZCQ) | 5 years
  ZCQ is a scale that measures physical function, symptom severity, and patient satisfaction for patients with spinal stenosis.
Quality of Life | 5 years
  Assessment of the patient's Quality of Life as measured by the Health Outcomes Survey and EQ-5D-5L
VAS Leg Pain | 5 years
  Change in the assessment of leg pain compared to pre-surgery as measured by a Visual Analog Scale (VAS) (on the 100mm scale).
VAS Back Pain | 5 years
  Change in the assessment of back pain compared to pre-surgery as measured by a Visual Analog Scale (VAS) (on the 100mm scale).

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - Center for Neurology and Spine, Phoenix, Arizona
  - Arizona Brain and Spine, Scottsdale, Arizona
  - Northwest NeuroSpecialists, Tucson, Arizona
  - The Spine Institute, Center for Spine Restoration, Santa Monica, California
  - Cantor Spine institute, Fort Lauderdale, Florida
  - Southeastern Integrated Medical, Gainesville, Florida
  - The Orthopaedic Institute, Gainesville, Florida
  - The BACK Center, Melbourne, Florida
  - All Florida Orthopaedics, St. Petersburg, Florida
  - Laser Spine Institute, Tampa, Florida
  - OrthoAtlanta, Lawrenceville, Georgia
  - Orthospine Center LTD, Palos Heights, Illinois
  - Orthopedic Center of Illinois, Springfield, Illinois
  - Brigham and Women's, Boston, Massachusetts
  - New England Orthopedic Surgeons, Springfield, Massachusetts
  - The Orthopedic Center of St. Louis, St Louis, Missouri
  - Orthopedic Sports Medicine & Spine Care Institute, St Louis, Missouri
  - North Jersey Brain and Spine Center, Oradell, New Jersey
  - IGEA Brain and Spine, Union, New Jersey
  - Spine and Orhtopedic Center of New Mexico, Roswell, New Mexico
  - Bassett Medical Center, Cooperstown, New York
  - Blue Ridge Bone and Joint, Arden, North Carolina
  - OrthoNeuro, Dublin, Ohio
  - Consulting Orthopaedic Associates, Sylvania, Ohio
  - OrthoTexas, Carrollton, Texas
  - Center for Spine Care, Dallas, Texas
  - NeoSpine, Seattle, Washington
  - Bighorn Medical Center, Cody, Wyoming